CLINICAL TRIAL: NCT04551404
Title: Transcranial Electrical and Acoustic Stimulation for Tinnitus: A Randomized Double Blind Clinical Trial
Brief Title: Transcranial Electrical and Acoustic Stimulation for Tinnitus
Acronym: tEAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: tEAS
Record Dates: First submitted 2020-08-09; First posted 2020-09-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Tinnitus; Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation; RNA, Transfer, Ser

STUDY DESIGN:
Intervention Model Description: The crossover within-person design with 2 groups, 2 active conditions and appropriate control/pseudo-placebo/sham session is double-blinded. Overall, participants will undergo 20 stimulation visits and 6 additional assessment visits.
  Prior to conducting the above study, a pilot study of 40 patients and just 6 visits will be conducted to validate clinical procedures and outcomes. This procedure was approved by the ethics committee.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Intervention(s) A (Experimental): TRNS bilateral temporal regions combined with AS for 20 minutes
  Sham-tRNS bilateral temporal regions combined with Sham-AS for 20 minutes
  Interventions: Other: transcranial Random Noise Stimulation (tRNS) with acoustic stimulation (AS)
- Study Intervention(s) B = Control Intervention (Experimental): TRNS bilateral temporal regions for 20 minutes
  Sham-tRNS bilateral temporal regions for 20 minutes
  Interventions: Other: transcranial Random Noise Stimulation (tRNS) without acoustic stimulation (AS)

INTERVENTIONS:
Other: transcranial Random Noise Stimulation (tRNS) with acoustic stimulation (AS) — The study intervention consists of a bilateral tRNS application over temporal regions, parallel to the application of AS with WN 15 dB above the individual MML in one study arm. TRNS will be applied using two electrodes (35 qcm, 0,9% saline -soaked). Stimulus intensity will be below individual sensation threshold, but max. 2 mA. AS will never surpass 85 dB SPL at the ears.
  Arms: Study Intervention(s) A
Other: transcranial Random Noise Stimulation (tRNS) without acoustic stimulation (AS) — The study intervention consists of a bilateral tRNS application over temporal regions
  Arms: Study Intervention(s) B = Control Intervention

SUMMARY:
Transcranial electrical stimulation (tES) is an umbrella term for non-invasive brain stimulation using weak currents. It comprises transcranial direct current stimulation (tDCS), which is the most established and used method applying constant direct current, transcranial alternating current stimulation (tACS) with sinusoidal current in a fixed frequency, and finally transcranial random noise stimulation (tRNS), which is a subform of tACS generating a random range of low and high frequency alternating currents.

A pilot study conducted by Shekhawat and colleagues in 2015 tested the effects of simultaneous electrical and acoustic stimulation. Using tDCS and bilateral broadband noise simultaneously, they found that more tinnitus patients report an improvement in tinnitus perception in comparison to conditions only using tDCS or sham. Further similar approaches very published in recent years, namely a pilot study conducted by Teissmann et al in 2014; study protocols of Rabau et al. in 2015 and Shekhawat et al. in 2015; and an experimental study by Lee et al. in 2017. Results were indicative of a superior efficacy of combined electrical and acoustic approaches, while large-scale controlled studies have not been performed. The need for extension and replication of these approaches is therefore timely.

The aim behind our proposed approach, similar to the bimodal approaches above, is to couple the effects of tRNS and acoustic stimulation (AS) for better temporary tinnitus suppression and possible reversal of maladaptive neuroplasticity related to tinnitus. We aim at targeting the (bilateral) auditory cortex with tRNS as in former studies and combine it with white noise (WN) stimulation. This specific combination is novel in its nature and is building on cortical excitability following tRNS.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years to 75 years of age (younger age limit according to corona virus protection concepts and measures of the FOPH: Schutzkonzepte und -massnahmen (admin.ch))
* Persistent chronic tinnitus with duration of more than 3 months
* Signed Informed Consent after being informed about the study
* Fluent in German or English
* Tinnitus with a THI Grade 2 to 4 (18-76 points)
* Willing and able to attend the study visits

Exclusion Criteria:

* Actual neurological or psychiatric disorders
* Hyperacusis
* Regular intake of medication influencing the central nervous system (e.g. neuroleptics, hypnotics, sedatives, and anti-epileptics)
* Implanted pacemaker
* Surgical implants in the head region, such as cochlea implants
* Asymmetrical hearing (more than 20dB side difference), pantonal hearing loss > 40dB in any measured frequency up to 2kHz
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Known or suspected non-compliance, drug or alcohol abuse
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Change of self-report Visual Analogue Scale (VAS) ratings on tinnitus severity (loudness, distress) | up to 6 months
  Minmum value = 1, maximum value =10. The higher scores means a worse outcome.
Change of minimum masking level (MML) | up to 6 months

SECONDARY OUTCOMES:
event-related EEG power in alpha band | up to 6 months
  The influence of simultaneous tRNS and AS stimulation on neurophysiology will be investigated as a secondary outcome. Resting state and event-related EEG (auditory oddball) (Attias et al., 1993) will be recorded for that purpose.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, University Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Antal A, Herrmann CS. Transcranial Alternating Current and Random Noise Stimulation: Possible Mechanisms. Neural Plast. 2016;2016:3616807. doi: 10.1155/2016/3616807. Epub 2016 May 3. PMID 27242932
- [Background] Claes L, Stamberger H, Van de Heyning P, De Ridder D, Vanneste S. Auditory cortex tACS and tRNS for tinnitus: single versus multiple sessions. Neural Plast. 2014;2014:436713. doi: 10.1155/2014/436713. Epub 2014 Dec 22. PMID 25587455
- [Background] Joos K, De Ridder D, Vanneste S. The differential effect of low- versus high-frequency random noise stimulation in the treatment of tinnitus. Exp Brain Res. 2015 May;233(5):1433-40. doi: 10.1007/s00221-015-4217-9. Epub 2015 Feb 19. PMID 25694243
- [Background] Kreuzer PM, Poeppl TB, Rupprecht R, Vielsmeier V, Lehner A, Langguth B, Schecklmann M. Daily high-frequency transcranial random noise stimulation of bilateral temporal cortex in chronic tinnitus - a pilot study. Sci Rep. 2019 Aug 22;9(1):12274. doi: 10.1038/s41598-019-48686-0. PMID 31439873
- [Background] Lee HY, Choi MS, Chang DS, Cho CS. Combined Bifrontal Transcranial Direct Current Stimulation and Tailor-Made Notched Music Training in Chronic Tinnitus. J Audiol Otol. 2017 Apr;21(1):22-27. doi: 10.7874/jao.2017.21.1.22. Epub 2017 Mar 30. PMID 28417104
- [Background] Mohsen S, Mahmoudian S, Talebian S, Pourbakht A. Prefrontal and auditory tRNS in sequence for treating chronic tinnitus: a modified multisite protocol. Brain Stimul. 2018 Sep-Oct;11(5):1177-1179. doi: 10.1016/j.brs.2018.04.018. Epub 2018 Apr 25. No abstract available. PMID 29730252
- [Background] Rabau S, Van Rompaey V, Van de Heyning P. The effect of Transcranial Direct Current Stimulation in addition to Tinnitus Retraining Therapy for treatment of chronic tinnitus patients: a study protocol for a double-blind controlled randomised trial. Trials. 2015 Nov 10;16:514. doi: 10.1186/s13063-015-1041-2. PMID 26554670
- [Background] Shekhawat GS, Kobayashi K, Searchfield GD. Methodology for studying the transient effects of transcranial direct current stimulation combined with auditory residual inhibition on tinnitus. J Neurosci Methods. 2015 Jan 15;239:28-33. doi: 10.1016/j.jneumeth.2014.09.025. Epub 2014 Oct 5. PMID 25285987
- [Background] Teismann H, Wollbrink A, Okamoto H, Schlaug G, Rudack C, Pantev C. Combining transcranial direct current stimulation and tailor-made notched music training to decrease tinnitus-related distress--a pilot study. PLoS One. 2014 Feb 25;9(2):e89904. doi: 10.1371/journal.pone.0089904. eCollection 2014. PMID 24587113
- [Background] Van Doren J, Langguth B, Schecklmann M. Electroencephalographic effects of transcranial random noise stimulation in the auditory cortex. Brain Stimul. 2014 Nov-Dec;7(6):807-12. doi: 10.1016/j.brs.2014.08.007. Epub 2014 Aug 26. PMID 25245591
- [Background] Vanneste S, Fregni F, De Ridder D. Head-to-Head Comparison of Transcranial Random Noise Stimulation, Transcranial AC Stimulation, and Transcranial DC Stimulation for Tinnitus. Front Psychiatry. 2013 Dec 18;4:158. doi: 10.3389/fpsyt.2013.00158. eCollection 2013. PMID 24391599
- [Derived] Martins ML, Kleinjung T, Meyer M, Raveenthiran V, Wellauer Z, Peter N, Neff P. Transcranial electric and acoustic stimulation for tinnitus: study protocol for a randomized double-blind controlled trial assessing the influence of combined transcranial random noise and acoustic stimulation on tinnitus loudness and distress. Trials. 2022 May 19;23(1):418. doi: 10.1186/s13063-022-06253-5. PMID 35590399